CLINICAL TRIAL: NCT01254734
Title: Outcomes in Transoral Robotic Microsurgery for Head and Neck Tumors
Brief Title: Transoral Robotic Surgery in Treating Patients With Benign or Stage I-IV Head and Neck Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study will be rewritten as a data registry study
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09206; NCI-2010-02169 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-11-03; First posted 2010-12-07 (Estimated); Last update posted 2014-11-10 (Estimated); Status verified 2014-11

CONDITIONS: Recurrent Adenoid Cystic Carcinoma of the Oral Cavity; Recurrent Lymphoepithelioma of the Nasopharynx; Recurrent Lymphoepithelioma of the Oropharynx; Recurrent Mucoepidermoid Carcinoma of the Oral Cavity; Recurrent Squamous Cell Carcinoma of the Hypopharynx; Recurrent Squamous Cell Carcinoma of the Larynx; Recurrent Squamous Cell Carcinoma of the Lip and Oral Cavity; Recurrent Squamous Cell Carcinoma of the Nasopharynx; Recurrent Squamous Cell Carcinoma of the Oropharynx; Recurrent Verrucous Carcinoma of the Larynx; Recurrent Verrucous Carcinoma of the Oral Cavity; Stage I Adenoid Cystic Carcinoma of the Oral Cavity; Stage I Lymphoepithelioma of the Nasopharynx; Stage I Lymphoepithelioma of the Oropharynx; Stage I Mucoepidermoid Carcinoma of the Oral Cavity; Stage I Squamous Cell Carcinoma of the Hypopharynx; Stage I Squamous Cell Carcinoma of the Larynx; Stage I Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage I Squamous Cell Carcinoma of the Nasopharynx; Stage I Squamous Cell Carcinoma of the Oropharynx; Stage I Verrucous Carcinoma of the Larynx; Stage I Verrucous Carcinoma of the Oral Cavity; Stage II Adenoid Cystic Carcinoma of the Oral Cavity; Stage II Lymphoepithelioma of the Nasopharynx; Stage II Lymphoepithelioma of the Oropharynx; Stage II Mucoepidermoid Carcinoma of the Oral Cavity; Stage II Squamous Cell Carcinoma of the Hypopharynx; Stage II Squamous Cell Carcinoma of the Larynx; Stage II Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage II Squamous Cell Carcinoma of the Nasopharynx; Stage II Squamous Cell Carcinoma of the Oropharynx; Stage II Verrucous Carcinoma of the Larynx; Stage II Verrucous Carcinoma of the Oral Cavity; Stage III Adenoid Cystic Carcinoma of the Oral Cavity; Stage III Lymphoepithelioma of the Nasopharynx; Stage III Lymphoepithelioma of the Oropharynx; Stage III Mucoepidermoid Carcinoma of the Oral Cavity; Stage III Squamous Cell Carcinoma of the Hypopharynx; Stage III Squamous Cell Carcinoma of the Larynx; Stage III Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage III Squamous Cell Carcinoma of the Nasopharynx; Stage III Squamous Cell Carcinoma of the Oropharynx; Stage III Verrucous Carcinoma of the Larynx; Stage III Verrucous Carcinoma of the Oral Cavity; Stage IV Adenoid Cystic Carcinoma of the Oral Cavity; Stage IV Lymphoepithelioma of the Nasopharynx; Stage IV Lymphoepithelioma of the Oropharynx; Stage IV Mucoepidermoid Carcinoma of the Oral Cavity; Stage IV Squamous Cell Carcinoma of the Hypopharynx; Stage IV Squamous Cell Carcinoma of the Larynx; Stage IV Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IV Squamous Cell Carcinoma of the Nasopharynx; Stage IV Squamous Cell Carcinoma of the Oropharynx; Stage IV Verrucous Carcinoma of the Larynx; Stage IV Verrucous Carcinoma of the Oral Cavity
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients undergo transoral robotic microsurgery.
  Interventions: Procedure: transoral robotic surgery; Other: laboratory biomarker analysis; Procedure: quality-of-life assessment

INTERVENTIONS:
Procedure: transoral robotic surgery — Undergo transoral robotic microsurgery
Other: laboratory biomarker analysis — Correlative studies
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment

SUMMARY:
RATIONALE: Transoral robotic surgery (TORS) is a less invasive type of surgery for head and neck cancer and may have fewer side effects and improve recovery. PURPOSE: This clinical trial studies how transoral robotic surgery works in treating patients with benign or stage I-IV head and neck cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES: To conduct a pilot study at City of Hope (COH) which assesses the feasibility and safety of TORS (Transoral robotic surgery), including: total operative time, blood loss, hospitalization time, need to convert to an open procedure, intra-operative as well as post-operative complications. SECONDARY OBJECTIVES: I. To collect data on oncologic outcomes, disease free survival, local control rate and overall survival. II. To collect normative data regarding objective functional outcomes (FO) which may impact quality of life in patients undergoing TORS, including need for adjunctive procedures, such as gastrostomy tube placement and tracheostomy placement, and with regards to speech, swallowing function and pain, using patient-report outcomes instruments. OUTLINE: Patients undergo transoral robotic microsurgery. After completion of study treatment, patients are followed up periodically for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients clinical, radiologic or pathologic evidence of a benign or malignant tumor in the oral cavity, oropharynx, nasopharynx, hypopharynx, larynx, retropharynx or parapharyngeal space
* Surgical access is amenable to treatment with conventional transoral surgical procedures
* ASA (American Society of Anesthesiologists) performance status (PS) of 1-4 or ECOG (Eastern Cooperative Oncology Group) PS 0-3, thereby including a population that stands to gain the most from a minimally invasive surgical approach
* Patients should have no serious acute infection
* Patients must sign a study-specific informed consent form

Exclusion Criteria:

* Evidence of distant metastases (below the clavicle) by clinical or radiographic measures
* ASA score > 4; ECOG PS score > 3
* Pregnancy (during first or 3rd trimester - due to risks of anesthesia)
* The presence of medical conditions which contraindicate general anesthesia
* Unexplained fever or untreated, active infection
* Inability to obtain exposure to allow performance of the planned transoral surgical procedure
* Proposed surgical site with history of prior treatment: radiation
* Tumor adherent to carotid artery or jugular vein
* Fixation to pre-vertebral tumor
* Mandibular invasion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2011-04; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Assessment of the feasibility of Transoral Robotic Surgery (TORS) in improving transoral accessibility within the upper aerodigestive tract in patients with benign or malignant head and neck tumors | From 6 months to 3 years after completion of study treatment
Assessment of the total operative time to perform transoral surgery using TORS in patients with benign or malignant head and neck tumors | From 6 months to 3 years after completion of study treatment
Assessment of blood loss during transoral surgery using TORS in patients with benign or malignant head and neck tumors | From 6 months to 3 years after completion of study treatment
Assessment of hospitalization time of in patients with benign or malignant head and neck tumors undergoing transoral surgery using TORS | From 6 months to 3 years after completion of study treatment
Assessment of the need to convert to an open procedure during transoral surgery using TORS in patients with benign or malignant head and neck tumors | From 6 months to 3 years after completion of study treatment
Assessment of complications of transoral surgery using TORS in patients with benign or malignant head and neck tumors | From 6 months to 3 years after completion of study treatment

SECONDARY OUTCOMES:
Collection of data on oncologic outcomes, disease free survival, local control rate and overall survival. | From 6 months to 3 years after completion of study treatment
Assessment of quality of life outcomes in patients undergoing TORS using patient-report outcomes instruments | From 6 months to 3 years after completion of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ellie Maghami, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States